CLINICAL TRIAL: NCT02942862
Title: Evaluation of New Histoprognostic Criteria in a Retrospective Study of Colon Cancers Operated at Amiens University Hospital
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0021
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Orcein staining — Prognostic value of venous emboli detected by orcein staining

SUMMARY:
Colon cancer is a very common cancer. Prognosis and adjuvant treatment depend on the pathological results. Histoprognostic new factors have recently been published by several authors, but their validity is still debated.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated on for colon adenocarcinoma between 2004 and 2009 at the University Hospital of Amiens

Exclusion Criteria:

* Non-operated patients
* Patients operated on before 2004 or after 2009
* Patients operated in another center
* The other histological types
* Vicinity of tumors invading the colon by contiguity
* Colic metastasis
* Patients whose blocks or blades were not found in the archives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated on for colon adenocarcinoma between 2004 and 2009 at the University Hospital of Amiens
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Denis CHATELAIN, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France